CLINICAL TRIAL: NCT00085930
Title: Administration of Peripheral Blood T-Cells and EBV Specific CTLs Transduced to Express GD-2 Specific Chimeric T Cell Receptors to Patients With Neuroblastoma
Brief Title: Blood T-Cells and EBV Specific CTLs Expressing GD-2 Specific Chimeric T Cell Receptors to Neuroblastoma Patients
Acronym: NESTLES
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13149-NESTLES; NESTLES (Other: BCM CAGT); NCT00609206 (obsolete NCT alias)
Record Dates: First submitted 2004-06-17; First posted 2004-06-21 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EBV specific CTLs w/out lymphodepletion (Experimental): Escalating doses of 14g2a.zeta chimeric receptor transduced autologous EBV specific cytotoxic T-lymphocytes (EBV-CTL) and 14g2a.zeta transduced autologous peripheral blood T-cells administered to patients with Neuroblastoma.
  Interventions: Biological: EBV specific CTLs

INTERVENTIONS:
Biological: EBV specific CTLs — CTLs: 2x10e7 cells/m2
  Other Names: 14g2a.zeta Chimeric Recep Transduc (EBV-CTL) w/o Lymphodepl

SUMMARY:
Patients have high-risk neuroblastoma, a form of cancer typically found in children. The patients previously participated in a gene transfer research study using special immune cells. This research study combines two different ways of fighting disease, antibodies and T cells. Antibodies are types of proteins that protect the body from bacterial and other infections. T cells, also called cytotoxic T lymphocytes or CTLs, are special infection-fighting blood cells that can kill some tumor cells. Both antibodies and T cells have been used to treat patients with cancers and while they have shown promise, they have not been strong enough to cure most patients. The antibody used in this study is called 14g2a. This antibody sticks to neuroblastoma cells because of a substance on the outside of these cells called GD2. 14g2a and other antibodies that bind to GD2 have been used to treat people with neuroblastoma. For this study 14g2a has been changed so that instead of floating free in the blood, it is now joined to T cells. When an antibody is joined to a T cell in this way it is called a chimeric receptor. T lymphocytes or CTLs can kill tumor cells but there normally are not enough of them to kill all tumor cells. Some researchers have taken T cells from a person's blood, grown more of them in the laboratory and then given them back to the patient. Sometimes an antibody or chimeric receptor is attached to these T cells to help them bind to tumor cells. These chimeric receptor-T cells seem to kill some of the tumor, but they don't last very long in the body and so the tumor eventually comes back. We have found that T cells that are also trained to recognize the virus that causes infectious mononucleosis, Epstein Barr Virus (EBV), can stay in the blood stream for many years. By joining the 14g2a antibody to the CTLs that recognize EBV, we believe we will make a cell that can last a long time in the body (because they are EBV-specific) and recognize and kill neuroblastoma cells (because an antibody that can recognize these cells has been placed on their surface). Patients received treatment with the immune cells described above. They may want to receive an additional dose of these cells. This is being offered as an option because their neuroblastoma has returned and they have enough cells remaining to provide the patients with an additional dose. These 14g2a antibody CTLs are an investigational product not approved by the Food and Drug Administration.

DETAILED DESCRIPTION:
Earlier, the patient gave us blood to make 14g2a chimeric receptor-T cells and 14g2a chimeric receptor-EBV CTLs in the laboratory. These cells were grown and frozen for the patient. The patient received treatment with these cells. However, there are enough cells remaining that we are able to offer to treat the patient with an additional dose if they would like.

As with the original treatment, the patient will be given an injection of cells into the vein through and IV. Before the injection is received, the patient will be given a dose of Benadryl and Tylenol. The injection will take about 2 minutes. We will follow the patient in the clinic after the injection for 3 hours. The treatment will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital.

Medical tests before treatment--

Before being treated, the patient will receive a series of standard medical tests:

* Physical exam
* Blood tests to measure blood cells, kidney and liver function
* Measurements of tumor by scans and bone marrow studies if the bone marrow may show evidence of disease

Medical tests during and after treatment:

The patient will receive standard medical tests when they are getting the infusions and after:

* Physical exams
* Blood tests to measure blood cells, kidney and liver function
* Measurements of tumor by scans and bone marrow studies if the bone marrow had evidence of disease 6 weeks after each infusion

Because the patient has received cells with a new gene in them the patient will be followed for a total of 15 years to see if there are any long term side effects of gene transfer. If they have a procedure related to their tumor (for example a biopsy or tumor resection), we will request permission to obtain a tissue sample. This will help investigators learn more about T cell and CTL treatment of neuroblastoma. In the event of death, we will request permission to perform an autopsy to learn more about the effects of these infusions on the disease.

ELIGIBILITY:
Inclusion Criteria:

High risk neuroblastoma with a history of persistent or relapsed disease, or after initial therapy

Patients must have a life expectancy of at least 12 weeks

Patients must have recovered from the toxic effects of all prior chemotherapy before entering this study

Patients must not be currently receiving any investigational agents or have not received any tumor vaccines within the previous 6 weeks

Patients must have an ANC > 500, platelet count > 20,000

Patients who have received prior therapy with murine antibodies must have documentation of absence of human anti-mouse antibodies (HAMA) prior to enrollment on this study

Patients must have bilirubin less than 3 times the upper limit of normal

Patients must have AST less than 5 times the upper limit of normal

Patients must have serum creatinine less than 3 times upper limit of normal

Patient may not have cardiomegaly or bilateral pulmonary infiltrates on chest radiograph. Patients may have pulmonary metastatic lesions

Patient may not have an oxygen requirement as defined by pulse oximetry of > 90% on room air

Patients must have Karnofsky score of > 60% if > 10 years old or Lansky performance score of greater than 60% if 10 years old or younger

Patients must have autologous transduced EBV-specific CTLs and transduced peripheral blood T-cells with 15% expression or greater of 14g2a.zeta determined by flow-cytometry

Sexually active patients must be willing to utilize one of the more effective birth control methods during the study and for 3 months after the study is concluded. The male partner should use a condom

Patients must not be pregnant or lactating

Patients must not have tumor in a location where enlargement could cause airway obstruction

Patients must not have a history of hypersensitivity to murine protein-containing products

Patients must not have a known sensitivity to rat monoclonal antibodies

Note: All labs must be collected within 10 days prior to initiation of study related treatment

Exclusion Criteria:

* Patients not meeting eligibility criteria

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2003-04; Primary Completion 2010-01 (Actual); Study Completion 2025-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of escalating doses of 14g2a.zeta chimeric receptor transduced autologous EBV specific cytotoxic T-lymphocytes (EBV-CTL) and 14g2a.zeta transduced autologous peripheral blood T-cells | 15 yrs
  Listings of adverse events by patients will include the time to onset, the duration of each event, the severity of each event, and the relationship of the event to study therapy, whether it was a serious event, and whether it caused withdrawal.

SECONDARY OUTCOMES:
Determine the differential survival and function of these two infused cell-types in vivo, in particular to determine if chimeric receptor transduced EBV-CTLs survive longer than transduced peripheral-blood T-cells. | 15 yrs
  To compare the in vivo survival and expansion of the T cells and the CTL and to determine if the T cells or the CTL expand more rapidly after infusion.
Determine anti-tumor effects of transduced peripheral blood T-cells and EBV specific CTLs in vivo. | 15 years
  Frequencies and proportions of anti-tumor activity based on evaluations of tumor size.
Compare the differential survival of these infused cells in an additional 6 patients treated at dose level #1 without CD45 antibody mediated lymphodepletion, to patients previously treated at dose levels #2 and #3. | 15 years
  Detect a 1-week half-life difference between dose level 1 and dose level 2

CONTACTS AND LOCATIONS:
Overall Officials: Helen E Heslop, MD, Study Director — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

REFERENCES:
- [Derived] Li CH, Sharma S, Heczey AA, Woods ML, Steffin DHM, Louis CU, Grilley BJ, Thakkar SG, Wu M, Wang T, Rooney CM, Brenner MK, Heslop HE. Long-term outcomes of GD2-directed CAR-T cell therapy in patients with neuroblastoma. Nat Med. 2025 Apr;31(4):1125-1129. doi: 10.1038/s41591-025-03513-0. Epub 2025 Feb 17. PMID 39962287
- [Derived] Louis CU, Savoldo B, Dotti G, Pule M, Yvon E, Myers GD, Rossig C, Russell HV, Diouf O, Liu E, Liu H, Wu MF, Gee AP, Mei Z, Rooney CM, Heslop HE, Brenner MK. Antitumor activity and long-term fate of chimeric antigen receptor-positive T cells in patients with neuroblastoma. Blood. 2011 Dec 1;118(23):6050-6. doi: 10.1182/blood-2011-05-354449. Epub 2011 Oct 7. PMID 21984804